CLINICAL TRIAL: NCT05099146
Title: Impact of Oral Health Educational Interventions on Oral Hygiene Status of Deaf Children - A Randomized Controlled Trial
Brief Title: Impact of Oral Health Education on Oral Hygiene Status of Deaf Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Maria Moin, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DowMDS
Record Dates: First submitted 2021-09-13; First posted 2021-10-29 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Motion Pictures; Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pictorial (Experimental): brushing technique taught by using pictures
  Interventions: Behavioral: pictures
- video (Experimental): brushing technique taught by showing video
  Interventions: Behavioral: video
- control (Experimental): only oral hygiene instructions provided
  Interventions: Behavioral: control

INTERVENTIONS:
Behavioral: pictures — pictures with brushing technique demonstrated technique for proper brushing
  Arms: pictorial
Behavioral: video — video of brushing technique demonstrated technique for proper brushing
  Arms: video
Behavioral: control — oral hygiene instructions provided
  Arms: control

SUMMARY:
Objective: To compare the impact of pictorial and video demonstration oral health educational interventions on oral hygiene status of children aged 12-16 years with hearing impairment.

Methods: This randomized controlled trial spanned over the period of three months was conducted in purposively selected three schools of deaf children of Karachi. Baseline dental examination was performed to assess the dental plaque and gingival status of study participants. Dental plaque and gingival status of the participants was assessed by employing the World Health Organization recommended Plaque Index and Gingival Index. The 60 children were than randomly allocated into three interventional groups, pictorial, video and control, 20 in each group. The children were examined again after one month of oral health education provision by single examiner. Tooth brushes were provided to students at the time of baseline examination to use for one month. Collected data was subjected to statistical analysis and described in terms of Mean and Standard Deviation, mixed model ANNOVA was applied to see the difference between the mean plaque and gingival scores of three groups after one month. The p-value of <0.05 was considered as statistically significant at the 95% confidence interval.

DETAILED DESCRIPTION:
Background: Health education, conventionally and appropriately, one of the foundation of preventive dentistry, has over the years involved in significant investments of time, power, human resources and funds. Children with impaired hearing have difficulties in speaking and communication and so learning process would be longer and even more challenging than the other children without such disabilities.

Objective: To compare the impact of pictorial and video demonstration oral health educational interventions on oral hygiene status of children aged 12-16 years with hearing impairment.

Methods: This randomized controlled trial spanned over the period of three months was conducted in purposively selected three schools of deaf children of Karachi. Baseline dental examination was performed to assess the dental plaque and gingival status of study participants. Dental plaque and gingival status of the participants was assessed by employing the World Health Organization recommended Plaque Index and Gingival Index. The 60 children were than randomly allocated into three interventional groups, pictorial, video and control, 20 in each group. The children were examined again after one month of oral health education provision by single examiner. Tooth brushes were provided to students at the time of baseline examination to use for one month. Collected data was subjected to statistical analysis and described in terms of Mean and Standard Deviation, mixed model ANNOVA was applied to see the difference between the mean plaque and gingival scores of three groups after one month. The p-value of <0.05 was considered as statistically significant at the 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Children with hearing impairment
* Children with age of 12-16 years
* Children with no systemic disease
* Children with Plaque adhering to the free gingival margin, more than one third and more than two thirds of tooth surface
* Children with mild, moderate and severe gingivitis
* Agreement on written accent
* Agreement to comply with study visits and procedure

Exclusion Criteria:

* Conditions requiring antibiotic pre-medication prior to dental examination
* Children with extensive dental calculus

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-10-05 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
change of dental plaque status | one month
  Assessed by plaque index, Change of plaque score From high to low levels after1 month

SECONDARY OUTCOMES:
Change in oral hygiene status | one month
  Assessed by oral hygiene index, Change of Oral hygiene scores From high to low levels after 1 month

CONTACTS AND LOCATIONS:
Overall Officials: MARIA MOIN, MDS, Principal Investigator — DOW UNIVERSITY OF HEALTH SCINCES
Locations (1):
- Ida Rieu College For Blind And Deaf, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No